CLINICAL TRIAL: NCT01190501
Title: Arterial Stiffness Index as a Predictor of Surgically Correctable Primary Aldosteronism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 07 326 03
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Adenoma
Keywords: blood pressure; antihypertensive treatments
MeSH Terms: conditions — Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- complier device (Experimental)
  Interventions: Device: complier device

INTERVENTIONS:
Device: complier device — The procedure of use of complier has to follow the recommendations for standardization of subject conditions.
  Assessment of arterial distensibility: pulse wave velocity (PWV), aortic stiffness is assessed by PWV which is a classic index of arterial stiffness. A semi-automatic device is used to measure carotid-femoral PWV. The distance covered by the pulse wave is measured on the surface of the body and represented the distance between the 2 recording sites.

SUMMARY:
Our main objective is to assess whether aortic stiffness is a predictor of blood pressure response after surgery in patients with an aldosterone producing adenoma or a unilateral adrenal hyperplasia.

DETAILED DESCRIPTION:
Secondary objectives are to investigate whether aortic stiffness predicts cardiovascular , operative and postoperative morbid-mortality at 1 year, to evaluate the benefit of adrenalectomy in patients with primary aldosteronism due to unilateral adrenal hyperplasia and in patients with aldosterone producing adenoma associated with controlateral adrenal morphological abnormalities, and to participate to a national DNA repository of patients with primary aldosteronism.

ELIGIBILITY:
Inclusion Criteria:

* patients with a surgically correctable primary aldosteronism due to an aldosterone producing adenoma or an unilateral adrenal hyperplasia
* primary aldosteronism demonstrated by hormonal essays
* hight resolution adrenal CT scan
* operative decision based on the usual criteria of the different referent centers

Exclusion Criteria:

* patient's refusal to undergo the surgery or to participate in the study
* the patients with PA due to bilateral adrenal hyperplasia or with idiopathic primary aldosteronism, and patients with a biochemical diagnosis of PA without evidence for a lateralized aldosterone excess.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-06; Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Responders to surgery, patients not receiving aldosterone antagonists, with mean-24h-ABP < 130/80 mmHg with or without antihypertensive treatment | 2 years

SECONDARY OUTCOMES:
Day-time and night-time ABP and circadian BP variability, number of antihypertensive agents at 1 year after surgery, prediction of post-operative complications, prediction of cardiovascular morbidity at 1 year. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chamontin, MD, Study Director — University Hospital, Toulouse; Pierre-François Plouin, MD, Principal Investigator — APHP-HEGP; Philippe Gosse, MD, Principal Investigator — University Hospital, Bordeaux; Jean-Philippe Baguet, MD, Principal Investigator — CHU Grenoble michalon; Pierre Lantelme, MD, Principal Investigator — Hospices de Lyon; Xavier Girerd, MD, Principal Investigator — APHP-Pitié Salpêtrière; Claire Mounier-Vehier, MD, Principal Investigator — CHR Lille; Yves Resnik, MD, Principal Investigator — CHU caen Côte de Nacre
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No